CLINICAL TRIAL: NCT05417581
Title: Mitochondrial Oxygraphy on Subcutaneous and Peri-visceral Adipose Tissue: Influence of Body Composition
Acronym: OxMiTiAd
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty of recruitment for Groups 1 and 3 not allowing all recruitment to be carried out over a reasonable period of time, it was decided to close this project
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: RBHP 2020 RICHARD; 2020-A03309-30 (Other: ANSM)
Record Dates: First submitted 2022-05-17; First posted 2022-06-14 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Digestive Organs--Cancer; Bariatric Surgery Candidate; Parietal Region Trauma
Keywords: Mitochondria; Oxygraphy; Adipose Tissue; Body Mass Index; Digestive surgery
MeSH Terms: conditions — Craniocerebral Trauma

STUDY DESIGN:
Intervention Model Description: all participants receive the same intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients (Experimental): a sample of adipose tissue will be collected during the scheduled surgery
  Interventions: Procedure: adipose surgery

INTERVENTIONS:
Procedure: adipose surgery — A quantity of adipose tissue equivalent to 10-20 cubic centimeter will be removed subcutaneously and from the omentum during surgical procedures (oncological, bariatric)

SUMMARY:
The objective of this study is to adapt the oxygraphy technique on human adipocytes and to characterize respiration measurements according to patients' body mass index and white adipose tissue localization (subcutaneous vs visceral).

DETAILED DESCRIPTION:
During digestive surgery: oncological and bariatric surgery, it is possible to collect a small volume of subcutaneous and epiplonic adipose tissue (10-20 cc). We wish to collect these samples in order to develop the technique of oxygenography on permeabilized adipocytes. In order to characterize these measurements, they will be related to the clinical data of the patients usually collected in the framework of the preoperative assessment including the body mass index (BMI). The measured adipocyte data will thus be normalized to three BMI classes: ≤ 20, > to 20 < 30, and ≥ to 30 kg∙m-2.

Primary end point is to validate the measurement of mitochondrial respiration under oxidophosphorylating conditions by determining indicators of the distribution of mitochondrial respiration values (mean, standard deviation, skewness, kurtosis, coefficient of variation) as a function of patients' body mass index.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing oncological, bariatric, parietal surgery
* Patients able to give an informed consent
* Patients affiliated to an Health Care insurance
* Patients aged over 18

Exclusion Criteria:

* Patients under guardianship, curatorship or deprived of freedom
* Pregnant or breastfeeding women
* Participation refusal
* Patients under chemotherapy
* Patients with peritonitis and infectious parietal processes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2023-04-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of mitochondrial respiration on adipose tissue by oxygraphy | day 1
  Mitochondrial respiration measurements in oxydophosphorylated conditions. For each patient measurements using ADP and carbohydrate or lipid substrates of the respiratory chain complexes for both the subcutaneous and the visceral tissue.

SECONDARY OUTCOMES:
mitochondrial respiration values depending on patients BMI by oxygraphy | day 1
  Identification of mitochondrial respiration discrimination factors
comparing mitochondrial respiration values depending on tissue location by oxygraphy | day 1
  Identification of mitochondrial respiration discrimination factors
comparing mitochondrial respiration values depending on anthropometric data by oxygraphy | day 1
  Identification of mitochondrial respiration discrimination factors

CONTACTS AND LOCATIONS:
Overall Officials: Ruddy RICHARD, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU clermont-ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Guerrier L, Bacoeur-Ouzillou O, Touron J, Mezher S, Cassagnes L, Vieille-Marchiset A, Chanon S, Pereira B, Pezet D, Pinel A, Gagniere J, Malpuech-Brugere C, Richard R. Mitochondrial respiration in white adipose tissue is dependent on body mass index and tissue location in patients undergoing oncological or parietal digestive surgery. FASEB J. 2025 Jan 31;39(2):e70350. doi: 10.1096/fj.202402243R. PMID 39856788